CLINICAL TRIAL: NCT00044837
Title: A Phase I, Pharmacokinetic Study of Hormone Replacement Therapy in HIV-1-Infected, Postmenopausal Women on Nelfinavir, Lopinavir/Ritonavir, or Efavirenz
Brief Title: Hormone Replacement Therapy and Anti-HIV Drugs in HIV-Infected, Postmenopausal Women
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Purpose: Treatment
Other Study IDs: ACTG A5119; AACTG A5119
Record Dates: First submitted 2002-09-05; First posted 2002-09-09 (Estimated); Last update posted 2015-06-04 (Estimated); Status verified 2003-06

CONDITIONS: HIV Infections
Keywords: Lopinavir; HIV-1; HIV Protease Inhibitors; Ritonavir; Postmenopause; Reverse Transcriptase Inhibitors; Pharmacokinetics; Area Under Curve; Hormone Replacement Therapy; efavirenz; estradiol
MeSH Terms: conditions — HIV Infections | interventions — Medroxyprogesterone Acetate; Estradiol

INTERVENTIONS:
Drug: Medroxyprogesterone acetate
Drug: Estradiol

SUMMARY:
The purpose of this study is to find out if the anti-HIV drugs nelfinavir (NFV), lopinavir/ritonavir (LPV/r), and efavirenz (EFV) change the amount of estrogen in the blood when taken along with hormone replacement therapy (HRT) for menopause.

HRT can be helpful for treating bothersome symptoms of menopause. However, it is not routinely used in HIV-infected postmenopausal women because it is not known how HRT interacts with anti-HIV drugs. The information obtained from this study will help doctors make recommendations for HRT in postmenopausal HIV-infected women.

DETAILED DESCRIPTION:
The benefits of hormone replacement therapy (HRT) in HIV-negative postmenopausal women include the abatement of menopausal symptoms such as hot flashes, insomnia, mood changes, vaginal dryness, urogenital and skin changes, and memory loss. HRT may also decrease risk for primary cardiovascular disease, osteoporosis, colon cancer, and possibly Alzheimer's disease and age-related macular degeneration. There may also be an overall survival benefit for HIV-negative postmenopausal women taking hormone replacement therapy. Despite the potential benefits of postmenopausal hormone replacement, it is seldom used in HIV-infected postmenopausal women. One concern about HRT in HIV-infected women is the potential for interaction with antiretroviral (ARV) drugs. Although the effect of HRT on ARV drug levels is likely to be small, it is important to evaluate the safety of administering HRT concurrently with ARVs. The information obtained from this study will help shape recommendations for postmenopausal HRT in HIV-infected women.

Patients are enrolled into 1 of 4 study arms based on their current oral ARV regimens. Arm A takes NFV plus nucleoside reverse transcriptase inhibitors (NRTIs). Arm B takes LPV/r plus NRTIs. Arm C takes EFV plus NRTIs. Arm D enrolls HIV-infected patients not on current ARVs, or who are taking NRTIs only (no protease inhibitors [PIs] or nonnucleoside reverse transcriptase inhibitors [NNRTIs]). All arms receive HRT with oral estradiol and medroxyprogesterone acetate for 12 weeks. Arms A, B, and C have intensive PI or NNRTI pharmacokinetic (PK) sampling at entry and Week 4. All arms have estradiol PK sampling at Week 4. Clinical and laboratory evaluations are done at entry, Week 4, and Week 12.

ARVs are not provided by this study. Only HRT is provided.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are postmenopausal women over 18 years old.
* Are infected with HIV.
* Have a CD4 cell count of 100 cells/mm3 or greater within 45 days prior to study entry.
* Have a plasma viral load less than 55,000 copies/ml within 45 days prior to study entry.
* Are willing to comply with study requirements. These include not changing smoking habits during the course of the study and not consuming caffeine or alcohol prior to PK sampling.
* Have had a Pap smear within 12 months prior to study entry.
* Meet one of the following requirements: a) patients must currently be on stable PI or EFV regimens plus 2 or more acceptable NRTIs, or b) patients must not currently be taking any ARVs, with the exception of an NRTI-only regimen.
* Have a way to obtain their ARVs outside of the study and agree to continue their ARV regimen for at least 12 weeks of the study.

Exclusion Criteria

Patients may not be eligible for this study if they:

* Have had breast or endometrial cancer, thrombophlebitis, or thromboembolism.
* Have had serious nausea, vomiting, or abdominal pain within 30 days prior to study entry.
* Have had a serious illness requiring systemic treatment and/or hospitalization within 14 days prior to study entry.
* Are allergic or sensitive to the drugs that will be used for HRT.
* Have undiagnosed postmenopausal bleeding.
* Have coronary artery disease.
* Have used hormonal therapies within 8 weeks prior to study entry.
* Have used DMPA (Depo Provera) within 180 days prior to study entry.
* Have used the anti-HIV drugs ZDV and d4T at the same time within 30 days prior to study entry.
* Have used other medications specified in the protocol within 30 days prior to study entry.
* Are using experimental drugs without the written approval of the study co-chairs.
* Are unable to adhere to the ARV or HRT medications while on study, in the opinion of the investigator.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120

CONTACTS AND LOCATIONS:
Overall Officials: Lori Kamemoto, Study Chair; Mary Vogler, Study Chair
Locations (1):
- Barbara Brizz, Rockville, Maryland, United States

REFERENCES:
- [Background] Clark RA, Cohn SE, Jarek C, Craven KS, Lyons C, Jacobson M, Kamemoto L. Perimenopausal symptomatology among HIV-infected women at least 40 years of age. J Acquir Immune Defic Syndr. 2000 Jan 1;23(1):99-100. doi: 10.1097/00126334-200001010-00016. No abstract available. PMID 10708064
- [Background] Gorski JC, Wang Z, Haehner-Daniels BD, Wrighton SA, Hall SD. The effect of hormone replacement therapy on CYP3A activity. Clin Pharmacol Ther. 2000 Oct;68(4):412-7. doi: 10.1067/mcp.2000.110560. PMID 11061581
- [Background] Porter VR, Greendale GA, Schocken M, Zhu X, Effros RB. Immune effects of hormone replacement therapy in post-menopausal women. Exp Gerontol. 2001 Feb;36(2):311-26. doi: 10.1016/s0531-5565(00)00195-9. PMID 11226745
- [Background] Ouellet D, Hsu A, Qian J, Locke CS, Eason CJ, Cavanaugh JH, Leonard JM, Granneman GR. Effect of ritonavir on the pharmacokinetics of ethinyl oestradiol in healthy female volunteers. Br J Clin Pharmacol. 1998 Aug;46(2):111-6. doi: 10.1046/j.1365-2125.1998.00749.x. PMID 9723818